CLINICAL TRIAL: NCT04275622
Title: The Effect of Lifestyle Intervention for Hypertriglyceridemia on the Pathogenesis of Adverse Pregnancy Outcome: the LITAPO Randomized Trial
Brief Title: The Effect of Lifestyle Intervention for Hypertriglyceridemia on the Pathogenesis of Adverse Pregnancy Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201906001RINC
Record Dates: First submitted 2020-02-09; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-11

CONDITIONS: Hypertriglyceridemia During Pregnancy
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group receives lifestyle intervention for hypertriglyceridemia.
  Interventions: Behavioral: Lifestyle including optimal exercise and diet modification.
- Control (No Intervention): Control group receives regular surveillance.

INTERVENTIONS:
Behavioral: Lifestyle including optimal exercise and diet modification. — The intervention group will receive diet education and be given exercise suggestion.
  Arms: Intervention

SUMMARY:
During pregnancy, hypertriglyceridemia is associated with adverse pregnancy outcomes, including gestational hypertension, preeclampsia, gestational diabetes mellitus, large for gestational age (LGA), and preterm delivery. However, whether lifestyle intervention for hypertriglyceridemia during pregnancy improves pregnancy outcomes remains unknown. Therefore, we will conduct a randomized controlled trial to investigate this issue.

At a tertiary medical center, we will enroll 70 pregnant women in this prospective, open-label, randomized controlled, pilot study comparing the effect of lifestyle intervention for hypertriglyceridemia versus control between Mar 2020 and Mar 2022. Pregnant women recruited will be randomized into two groups. The intervention group will receive lifestyle intervention; whereas the control group will receive regular surveillance only. Only intervention group will have diet education and exercise goal. They will go to dietitian OPD twice at GA 30-31+6 and 33-34+6 for Mediterranean diet education. As for exercise, participants in intervention group are asked to at least take 10000 steps 3 days a week. Diet modification and exercise intervention will persistent until delivery.

The primary end point is the change of biomarkers of preeclampsia and macrosomia, including maternal blood PlGF and sFLT1, and cord blood c-peptide, leptin, IGF-1, IGF-2, IGF-BP1 and IGF-BP3. The secondary end points include the change of frequency of adverse pregnancy outcomes, including individual outcome and the composite outcome, such as gestational hypertension, preeclampsia, preterm delivery, and large for gestational age (defined as birth weight ≥ 90th percentile), change of maternal body weight, change of maternal blood pressure, which is defined as 3 mm-Hg, change of maternal HOMA2-IR, change of maternal plasma triglyceride level and other lipid profile (total cholesterol, HDL, and LDL), echography finding of fetus, neonatal birth weight, change of glucose, and lipid profile (total cholesterol, HDL, LDL, and TG) of fetus cord blood, placental expression of preeclampsia (PlGF, sFLT1) and growth factors (IGF-1, 2, BP1 and BP3).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women older than 20-year-old
* During GA 24-28+6 weeks
* Carrying a singleton
* Having hypertriglyceridemia (plasma triglyceride at GA 24-28+6 excess 246 mg/dL but not higher than 1000 mg/dL).

Exclusion Criteria:

* Using steroid
* Using anti-platelet or anti-coagulant
* Using lipid-lowering agents
* Hypertriglyceridemia is caused by secondary cause, such as hypothyroidism, cushing syndrome, nephrotic syndrome, alcohol use or medication use.
* Have been diagnosed with chronic hypertension, overt diabetes mellitus, gestational diabetes mellitus, secondary hypertriglyceridemia, autoimmune disease, or malignancy.
* Have received the artificial fertilization.
* Not having fetus echography examination at GA 22-23+6
* Not going to deliver the baby at National Taiwan University Hospital
* Have underwent other clinical trials

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of biomarkers of preeclampsia | Through study completion, an average of 2 year
  including maternal blood PlGF (pg/mL) and sFLT1 (pg/mL)
Change of biomarkers of macrosomia | Through study completion, an average of 2 year
  such as cord blood c-peptide (μg/L)
Change of biomarkers of macrosomia | Through study completion, an average of 2 year
  such as cord blood leptin (ng/mL)
Change of biomarkers of macrosomia | Through study completion, an average of 2 year
  such as cord blood IGF-1 (ng/mL), IGF-2 (ng/mL)
Change of biomarkers of macrosomia | Through study completion, an average of 2 year
  such as cord blood IGF-BP1 (μg/mL), and IGF-BP3 (μg/mL)

SECONDARY OUTCOMES:
Change of frequency of adverse pregnancy outcomes, including individual outcome and the composite outcome | Through study completion, an average of 2 year
  such as gestational hypertension, preeclampsia, preterm delivery, and large for gestational age
Change of maternal body weight | Through study completion, an average of 2 year
  Maternal body weight change (kilograms)
Change of maternal plasma triglyceride level (mg/dL) and other lipid profile (total cholesterol, HDL, and LDL) | Through study completion, an average of 2 year
  Other lipid profile including total cholesterol (mg/dL), HDL (mg/dL), and LDL (mg/dL)
Change of maternal blood pressure | Through study completion, an average of 2 year
  which is defined as 3 mm-Hg
Change of maternal homeostatic model assessment 2 insulin resistance indexes (HOMA2-IR) | Through study completion, an average of 2 year
  Maternal HOMA2-IR change. The higher level of HOMA2-IR means the higher risk for insulin resistance.
Change of glucose level of fetus cord blood | Through study completion, an average of 2 year
  Change of glucose level (mg/dL) of fetus cord blood
Change of lipid profile of fetus cord blood | Through study completion, an average of 2 year
  including TG (mg/dL), total cholesterol (mg/dL), HDL (mg/dL), and LDL (mg/dL)
Echography finding of fetus | Through study completion, an average of 2 year
  including biparietal diameter (mm), femur length (mm), head circumference (mm), and abdominal circumference (mm)
Echography finding of fetus | Through study completion, an average of 2 year
  including estimated fetal weight (gm)
Neonatal birth weight | Through study completion, an average of 2 year
  Neonatal birth weight (grams)
Placental protein expression (immunohistochemistry or western blot) of preeclampsia biomarkers | Through study completion, an average of 2 year
  including PlGF and sFLT1
Placental protein expression (immunohistochemistry or western blot) of growth factors | Through study completion, an average of 2 year
  including IGF-1, IGF-2, IGF-BP1, and IGF-BP3

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan